CLINICAL TRIAL: NCT01143688
Title: Characterization of Placebo Responses in Stable Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Wechsler, MD, Michael Wechsler, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005P-002045; R21AT002793-01 (NIH); K24AT004095 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma Placebo Effects
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- albuterol inhaler (Active Comparator): albuterol
  Interventions: Drug: albuterol
- placebo inhaler (Placebo Comparator): placebo
  Interventions: Drug: placebo inhaler
- placebo acupuncture (Placebo Comparator): placebo
  Interventions: Procedure: placebo acupuncture

INTERVENTIONS:
Drug: albuterol
  Arms: albuterol inhaler
Drug: placebo inhaler
  Arms: placebo inhaler
Procedure: placebo acupuncture
  Arms: placebo acupuncture

SUMMARY:
The investigators hypothesize that different placebos will have different effects on subjective and objective asthma outcomes compared with actual therapy and natural history. .

Subjects with asthma are randomly treated with placebo inhaler, placebo acupuncture, albuterol inhaler, or "no treatment" in random order, on three different occasions each. At each of the 12 visits, spirometry is performed repeatedly over 2 hours. Maximum FEV1 achieved and an 11-point, self-reported scale of improvement are examined.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled asthma

Exclusion Criteria:

* no bronchodilator response

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wechsler, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 patients completed questionnaires, 46 patients had reversibility and were randomized, and 39 completed the whole trial. The data was solely based on the 39 subjects who completed the entire trial.
Groups:
- All Study Participants: Each study participant was randomized to a specific random sequence of interventions for visits 1-4 (e.g. first inhaled bronchodilator, then inhaled placebo, then sham acupuncture, then no intervention administered 3-7 days apart, or first sham acupuncture, then inhaled bronchodilator, then no intervention, then inhaled placebo administered 3-7 days apart, or any other combination of these four interventions in any order). This process was repeated for visits 5-8 and again for visits 9-12.
Period: Overall Study
Arm/Group | All Study Participants
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 28
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1
Description: The baseline FEV1 (before treatment) was subtracted from the maximum FEV1 recorded during the 2 h period following treatment. This difference value was then converted into percent improvement by dividing by baseline FEV1 and multiplying by 100. Each treatment was given 3 times to each patient, so we averaged the 3 values to yield the mean percent change in FEV1 for each condition.
Time Frame: FEV1 was assessed every 20 minutes for 2 hours at each visit. There were 4 visits in each block each visit separated by 3-7 days. There were three blocks each block separated by 3-7 days.
Population: Each patient went through each treatment arm (albuterol, placebo inhaler, placebo acupuncture, and no-intervention) once in block 1, then again in block 2, and again in block 3, for a total of 12 interventions of the course of the study.
Measure: Mean (Standard Error); unit: percentage change in FEV1
Groups:
- Albuterol Inhaler: Subjects will perform baseline spirometry. Subsequently subjects will be shown an unmarked metered-dose inhaler device. This inhaler contains active albuterol (90 mcg/puff). The subjects will be reminded that this inhaler may contain either albuterol or placebo, and will complete questionnaires documenting their expectations for improvement in lung function with this treatment. Subsequently subjects will inhale 4 puffs (360 mcg) of albuterol administered from this inhaler via a spacing device.
  Spirometry will be obtained every 20 minutes post inhalation and the maximal FEV1 measured over the subsequent 120 minutes will be recorded as the post-intervention response on that visit. In the time period between spirometry, subjects will sit quietly in a separate waiting area.
- Placebo Inhaler: Subjects will be shown an unmarked metered-dose inhaler similar to that used for bronchodilator testing. This placebo inhaler contains only propellant and inert ingredients (trichlorofluoromethane and dichlorodifluoromethane with lecithin). The subjects will be reminded that this inhaler may contain either albuterol or placebo. They will then inhale 4 puffs of the placebo inhaler containing only the propellant vehicle through a spacer. Spirometry will be obtained every 20 minutes post inhalation and the maximal FEV1 measured over the subsequent 120 minutes will be recorded as the post-intervention response on that visit. In the time period between spirometry, subjects will sit quietly in a separate waiting area.
- Placebo Acupuncture: Subjects will be instructed that they will receive one of three different acupuncture point combinations that may or may not be effective for asthma. Placebo acupuncture will be performed with a validated acupuncture device that allows patients to see an acupuncture needle enter their skin and actually feel the sensation of penetration. The needle penetrates up the needle shaft and never penetrates the point. The needle has been validated and shown to be indistinguishable from real acupuncture.
- No-intervention Control: Subjects will be instructed that they will receive no interventions on this visit.
  Spirometry will be obtained every 20 minutes for maximal FEV1 for 120 minutes. In the time period between spirometry, subjects will sit quietly in a separate waiting area.
Arm/Group | Albuterol Inhaler | Placebo Inhaler | Placebo Acupuncture | No-intervention Control
Number analyzed (Participants) | 39 | 39 | 39 | 39
percentage change in FEV1 | 20.1 (1.6) | 7.5 (1.0) | 7.3 (0.8) | 7.1 (0.8)

2. Secondary Outcome: Asthma Symptoms
Description: Subjective change in asthma symptoms on a visual-analogue scale with scores ranging from 0 (no positive change) to 10 (complete positive change). These subjective responses were then converted to percent change during the 2 hours by multiplying each score by 10. Each of these individual subject scores were then averaged to produce an average percent change in symptoms.
Time Frame: Assesed over 2 hours during each visit. There were 4 visits in each block each visit separated by 3-7 days. There were three blocks each block separated by 3-7 days.
Measure: Mean (Standard Error); unit: percent change in symptoms
Arm/Group | Albuterol Inhaler | Placebo Inhaler | Placebo Acupuncture | No-intervention Control
Number analyzed (Participants) | 39 | 39 | 39 | 39
percent change in symptoms | 50 (3.75) | 45 (3.75) | 46 (3.75) | 21 (3.45)

ADVERSE EVENTS:
Arm/Group | Albuterol Inhaler | Placebo Inhaler | Placebo Acupuncture | No-intervention Control
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39

LIMITATIONS AND CAVEATS:
The subjective scale did not encompass worsening of symptoms. Only studied acute asthmatic response, not chronic. Used single objective measure (FEV1) and single subjective measure. Did not assess subjective symptoms before each visit's intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No